CLINICAL TRIAL: NCT04513340
Title: AN OPEN LABEL, BALANCED, RANDOMISED, FOUR-TREATMENT, FOUR-PERIOD, FOUR-SEQUENCE, SINGLE INTRA-ORAL AND ORAL DOSE, CROSSOVER PHARMACOKINETICS STUDY OF WD-1603 EXTENDED-RELEASE CARBIDOPA/LEVODOPA TABLETS 25/100MG IN NORMAL, HEALTHY, ADULT HUMAN SUBJECTS UNDER FASTING AND FED CONDITIONS
Brief Title: WD-1603 PK Study Under Fasting and Fed Conditions in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong WD Pharmaceutical Co., Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WD-1603-1002
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): Treatment A will be given under fed conditions by intra-oral single dose administration
  Interventions: Drug: WD-1603 CARBIDOPA and LEVODOPA EXTENDED-RELEASE TABLETS
- Treatment B (Experimental): Treatment B will be given intra-orally and orally under fed conditions by single dose administration
  Interventions: Drug: WD-1603 CARBIDOPA and LEVODOPA EXTENDED-RELEASE TABLETS
- Treatment C (Experimental): Treatment C will be given orally under fed conditions by single dose administration
  Interventions: Drug: WD-1603 CARBIDOPA and LEVODOPA EXTENDED-RELEASE TABLETS
- Treatment D (Experimental): Treatment D will be given orally under fasting conditions by single dose administration
  Interventions: Drug: WD-1603 CARBIDOPA and LEVODOPA EXTENDED-RELEASE TABLETS

INTERVENTIONS:
Drug: WD-1603 CARBIDOPA and LEVODOPA EXTENDED-RELEASE TABLETS — CARBIDOPA and LEVODOPA EXTENDED-RELEASE TABLETS 25/100MG

SUMMARY:
The Phase 1 PK study is planned to evaluate the food effect on WD-1603 pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy adult human volunteers between 18 to 45 years of age (both inclusive).
2. Having a Body Mass Index (BMI) between 18.5 to 29.9 (both inclusive), calculated as weight in kg / height in m2.
3. Not having any significant disease or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12- lead ECG and X-ray chest (P/A view) recordings.
4. Able to understand and comply with the study procedures, in the opinion of the principal investigator.
5. Able to give voluntary written informed consent for participation in the trial.
6. In case of female subjects:

a. Surgically sterilized at least 6 months prior to study participation or If of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.

And b. Serum Pregnancy test must be negative.

Exclusion Criteria:

1. Known hypersensitivity or idiosyncratic reaction to Carbidopa or Levodopa or any of the excipients or any related drug.
2. History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
3. Ingestion of a medicine (prescribed & over the counter (OTC) medication including herbal remedies) at any time within 14 days before dosing in Period I. In any such case subject selection will be at the discretion of the Principal Investigator.
4. Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAIDs induced urticaria.
5. Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
6. A recent history of harmful use of alcohol (less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 ml of beer or 150 ml of wine or 45 ml of 40% distilled spirits, such as rum, whisky, brandy etc) or consumption of alcohol or alcoholic products within 48 hours prior to dosing in Period I.
7. Smokers, who smoke 10 or more than 10 cigarettes / day or inability to abstain from smoking during the study.
8. The presence of clinically significant abnormal laboratory values during screening.
9. History or presence of psychiatric disorders.
10. A history of difficulty in donating blood.
11. Donation of blood (1 unit or 350 mL) within a period of 90 days prior to the first dose of study medication.
12. Receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication**.

    ** If investigational medicinal product is received within 90 days where there is no blood loss except safety lab testing, subject can be included considering 10 half-lives duration of investigational medicinal product received.
13. A positive hepatitis screen including hepatitis B surface antigen and/or HCV antibodies.
14. A positive test result for HIV (1 &/or 2) antibody.
15. An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study medicine in period I. In any such case subject selection will be at the discretion of the Principal Investigator.
16. Consumption of grapefruit or grapefruit products within 72 hours prior to dosing in period-I.
17. Difficulty in swallowing oral solid dosage form like tablets or capsules.
18. Nursing mothers (females).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2020-09-05 (Estimated); Study Completion 2021-02-13 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day 1 and Day 2
  Pharmacokinetics Measurements to Determine Cmax for Carbidopa (CD) and Levodopa (LD) Plasma Concentrations
AUC0-t | Day 1 and Day 2
  Pharmacokinetics Measurements to Determine AUC0-t for Carbidopa (CD) and Levodopa (LD) Plasma Concentrations
AUC0-∞ | Day 1 and Day 2
  Pharmacokinetics Measurements to Determine AUC0-∞ for Carbidopa (CD) and Levodopa (LD) Plasma Concentrations

SECONDARY OUTCOMES:
Tmax | Day 1 and Day 2
  Pharmacokinetics Measurements to Determine Tmax for Carbidopa (CD) and
t1/2 | Day 1 and Day 2
  Pharmacokinetics Measurements to Determine t1/2 for Carbidopa (CD) and

CONTACTS AND LOCATIONS:
Locations (1):
- Lambda Therapeutic Research Ltd., Ahmedabad, India